CLINICAL TRIAL: NCT06687369
Title: Randomized, Multicenter, Multinational, Double-Blind Study to Compare the Pharmacokinetics, Efficacy, Safety and Immunogenicity of MB12 (Proposed Pembrolizumab Biosimilar) Versus Keytruda® in Combination With Chemotherapy for the Treatment of Patients With Advanced Stage IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC) (BENITO Study)
Brief Title: A Study to Compare Pharmacokinetics, Efficacy, Safety, and Immunogenicity of MB12 (Proposed Pembrolizumab Biosimilar) to Keytruda® in Non-small Cell Lung Cancer (BENITO Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB12-C-02-24
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non Squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB12 (Proposed Pembrolizumab Biosimilar) (Experimental): MB12 (Proposed Pembrolizumab Biosimilar) + Pemetrexed + Carboplatin/ Cisplatin
  Interventions: Drug: MB12 (Proposed Pembrolizumab Biosimilar); Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin
- EU- sourced Keytruda® (Active Comparator): EU- sourced Keytruda® + Pemetrexed + Carboplatin/ Cisplatin
  Interventions: Drug: EU-sourced Keytruda®; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin
- US- sourced Keytruda® (Active Comparator): US- sourced Keytruda® + Pemetrexed + Carboplatin/ Cisplatin
  Interventions: Drug: US-sourced Keytruda®; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: MB12 (Proposed Pembrolizumab Biosimilar) — 200mg IV, every 3 weeks on Day 1
  Arms: MB12 (Proposed Pembrolizumab Biosimilar)
Drug: EU-sourced Keytruda® — 200mg IV, every 3 weeks on Day 1
  Arms: EU- sourced Keytruda®
Drug: US-sourced Keytruda® — 200mg IV, every 3 weeks on Day 1
  Arms: US- sourced Keytruda®
Drug: Pemetrexed — 500 mg/m2 IV, every 3 weeks on Day 1
Drug: Carboplatin — Area under the curve (AUC) 5 IV, every 3 weeks on Day 1 for 4 cycles.
Drug: Cisplatin — 75 mg/m2 IV, every 3 weeks on Day 1 for 4 cycles

SUMMARY:
This is a randomized, multicenter, multinational, double-blind, integrated pharmacokinetics (PK) and efficacy similarity study to compare the PK, efficacy, safety, and immunogenicity of MB12 versus Keytruda® in combination with pemetrexed-platinum chemotherapy as first-line treatment in patients with metastatic non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female patients ≥18 years old at the time of signing the informed consent form (ICF).
2. Histologic or cytologic diagnosis of advanced NSCLC, stage IV (defined by the 8th edition of the Tumor Node Metastasis [TNM] classification), with no EGFR sensitizing (activating) mutation or ALK translocation, and who have not received prior systemic treatment for metastatic NSCLC. In those patients in whom the pleural or pericardial effusion is the only location of metastatic disease, confirmation of its malignant etiology is required.
3. At least 1 radiographically measurable lesion according to response evaluation criteria in solid tumors (RECIST) 1.1.
4. Known status of PD-L1 expression.
5. Performance based on the Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
6. Adequate hepatic, renal, hematologic, endocrine, and coagulation function.

Exclusion Criteria:

1. Predominantly squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the patient is not eligible.
2. Known history of central nervous system metastases and/or carcinomatous meningitis.
3. Prior anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T lymphocyte associated protein (CTLA)-4 therapy (including ipilimumab or any other antibody or drug that specifically targets co-stimulation of T-cells or immune checkpoints).
4. Major surgery within 3 weeks of the first dose of study treatment.
5. Active autoimmune disease that has required systemic treatment in the last 2 years.
6. Contraindication and/or intolerance to the administration of pembrolizumab or known sensitivity to any component of pembrolizumab.
7. Has a known sensitivity to any component of cisplatin, carboplatin, or pemetrexed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the pharmacokinetic (PK) bioequivalence of MB12, EU-sourced Keytruda® and US-sourced Keytruda® in combination with chemotherapy | Week 1 - Week 24
  Area under the concentration-time curve (AUC) between Cycle 1 and Cycle 2 (AUC from time 0 to 504 hours postdose [AUC0-504]. AUC at steady state (AUCss) between Cycle 7 and Cycle 8.
To demonstrate the efficacy equivalence of MB12 and Keytruda® in combination with chemotherapy administered as first-line treatment in patients with advanced/metastatic non-squamous NSCLC (any PD-L1 expression type). | Week 1 - Week 24
  Objective response rate (ORR), up to and including 24 weeks (end of Cycle 8)

SECONDARY OUTCOMES:
To assess the efficacy of MB12 as compared with Keytruda® based on other efficacy parameters and timepoints over the study period. | Week 1 - Week 52
  Objective response rate (ORR), Progression-free survival (PFS), Duration of response (DOR) and Overall survival (OS)
To compare the PK profile based on other PK parameters and timepoints (not covered by the primary PK endpoints) of MB12 as compared with Keytruda® over the study period. | Week 1 - Week 52
  Maximum concentration (Cmax), Time to maximum concentration (Tmax), Minimum concentration (Ctrough), Clearance (CL), Elimination half-life (t1/2), Distribution volume (Vd)
To assess the safety and tolerability of MB12 as compared with Keytruda® | Week 1 - Week 52
  Treatment-emergent adverse events (TEAEs)
To assess the immunogenicity of MB12 as compared with Keytruda® | Week 1 - Week 52
  Anti-drug antibodies (ADAs) and Neutralizing antibodies (NAbs) in ADA-positive samples

CONTACTS AND LOCATIONS:
Locations (80):
- Armenia (4):
  - Site 101001, Yerevan
  - Site 101002, Yerevan
  - Site 101003, Yerevan
  - Site 101004, Yerevan
- Bosnia and Herzegovina (3):
  - Site 103001, Sarajevo
  - Site 103002, Tuzla
  - Site 103003, Zenica
- Georgia (11):
  - Site 108004, Batumi
  - Site 108005, Kutaisi
  - Site 108011, Marneuli
  - Site 108001, Tbilisi
  - Site 108002, Tbilisi
  - Site 108003, Tbilisi
  - Site 108006, Tbilisi
  - Site 108007, Tbilisi
  - Site 108008, Tbilisi
  - Site 108009, Tbilisi
  - Site 108010, Tbilisi
- Japan (4):
  - Site 207002, Hakodate-shi
  - Site 207012, Okayama
  - Site 207010, Shinagawa-Ku
  - Site 207001, Shizuoka
- Jordan (7):
  - Site 114001, Amman
  - Site 114002, Amman
  - Site 114003, Amman
  - Site 114004, Amman
  - Site 114005, Amman
  - Site 114007, Amman
  - Site 114006, Irbid
- Malaysia (3):
  - Site 202001, Cheras
  - Site 202002, Kota Bharu
  - Site 202003, Kuala Selangor
- Research site 116001, Chisinau, Moldova
- Panama (3):
  - Site 304001, Panama City
  - Site 304002, Panama City
  - Site 304003, Panama City
- Poland (5):
  - Site 118004, Katowice
  - Site 118001, Lodz
  - Site 118005, Lublin
  - Site 118002, Prabuty
  - Site 118003, Słupsk
- Portugal (3):
  - Site 119001, Lisbon
  - Site 119002, Matosinhos Municipality
  - Site 119003, Porto
- Romania (5):
  - Site 120001, Cluj-Napoca
  - Site 120003, Craiova
  - Site 120004, Craiova
  - Site 120006, Floreşti
  - Site 120005, Timișoara
- Serbia (5):
  - Site 121001, Belgrade
  - Site 121002, Belgrade
  - Site 121004, Kamenitz
  - Site 121003, Kragujevac
  - Site 121005, Užice
- Slovakia (3):
  - Site 122003, Bardejov
  - Site 122001, Bratislava
  - Site 122002, Partizánske
- Spain (11):
  - Site 124006, A Coruña
  - Site 124013, Barcelona
  - Site 124011, Madrid
  - Site 124012, Madrid
  - Site 124008, Málaga
  - Site 124016, Murcia
  - Site 124003, Oviedo
  - Site 124001, Palma de Mallorca
  - Site 124014, Pontevedra
  - Site 124010, Santiago de Compostela
  - Site 124015, Valencia
- Thailand (7):
  - Site 206004, Bangkok
  - Site 206005, Bangkok
  - Site 206001, Chiang Mai
  - Site 206007, Chiang Rai
  - Site 206003, Khon Kaen
  - Site 206002, Nakhon Nayok
  - Site 206006, Songkhla
- Tunisia (5):
  - Site 112002, Aryanah
  - Site 112003, Aryanah
  - Site 112004, Aryanah
  - Site 112001, Sfax
  - Site 112005, Tunis